CLINICAL TRIAL: NCT05900830
Title: Effect of a Physical and Occupational Therapy Program on Academic Skills in Egyptian Children With Intellectual Disability
Brief Title: Therapy Program for Academic Skills in Children With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tayseer Saber Abdeldayem, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004233
Record Dates: First submitted 2023-02-10; First posted 2023-06-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Intellectual Disability, Mild; Educational Problems
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular | interventions — Play Therapy; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Quasi experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- common educational methods (Active Comparator): this group will receive common educational methods
  Interventions: Other: common educational methods
- play based program (Experimental): this group will get the combined selected physical and occupational therapy program
  Interventions: Other: play therapy

INTERVENTIONS:
Other: play therapy — A combined program based on physical and occupational therapy techniques within a play context
  Other Names: physical and occupational therapy program
  Arms: play based program
Other: common educational methods — the child will receive his education in a passive manner
  Other Names: Passive class room education
  Arms: common educational methods

SUMMARY:
The aim of this study is to investigate the effect of a physical and occupational therapy program on academic skills in a sample of Egyptian children with intellectual disability. It also aims to provide a program based on physical and occupational therapy activities and techniques to develop children's basic abilities through play to make learning more enjoyable

DETAILED DESCRIPTION:
This study hypothesis

1. There are statistically significant differences between the mean scores of the children of the experimental group in the pre and post measurements on the academic skills scale for children with mental disabilities and its sub-components in favor of the post measurement.
2. There are no statistically significant differences between the mean scores of the children of the experimental group in the post and follow-up measurements on the academic skills scale for children with mental disabilities and its sub-components.

RESEARCH QUESTION:

What is the effect of a physical and occupational therapy program in improving academic skills (reading - writing - arithmetic) in a sample of children with mild intellectual disabilities? The study should include 20 children diagnosed with mild intellectual disability according to Stanford Binet scale 5th edition between the age of 8 to 10 years old from both sexes recruited from Noor Al-Sabah Association for the Care and Rehabilitation of People with Intellectual Disabilities from children with mild mental disabilities

ELIGIBILITY:
Inclusion Criteria:

1. The child should be between 8 and 10 years of age of both sexes
2. The child should be of mild intellectual disabilities according to Stanford Binet scale 5th edition
3. The child should not be suffering from any apparent physical deformity in upper limbs, lower limbs or spine
4. The child should not suffer from any visual or auditory disorder

Exclusion Criteria:

1. Children out of age range
2. Children with moderate or severe intellectual disabilities
3. Children with physical deformities in upper limb, lower limb or spine
4. Children suffering from visual or auditory disorders
5. Children of parents who refuse to sign the consent form

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
The Academic Skills Scale for Children with Mild Intellectual Disabilities. | 2 months
  Reading and writing words, reading and writing simple sentences, knowledge of reading phenomena, comprehension., Reading, reading expression, reading and writing numbers and numbers, order and sequence, classification, relationships, arithmetic operations

SECONDARY OUTCOMES:
The Stanford-Binet Scale, the fifth edition | 2 months
  the Stanford-Binet Intelligence Scale Fifth Edition

CONTACTS AND LOCATIONS:
Overall Officials: Zienab M Mahmoud, PhD, Study Chair — Beni-Suef University; Nahed MG Makary, PhD, Study Chair — Beni-Suef University
Locations (1):
- Tayseer Younes, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
no personal data will be shared